CLINICAL TRIAL: NCT01694212
Title: Effect of Perioperative Topical Diclofenac on Intraocular Inflammation After Cataract Surgery and the Incidence of Postoperative Macular Edema in Patients With Diabetic Retinopathy
Brief Title: Preoperative Topic Diclofenac as a Prevention of Postoperative Macular Edema in Patients With Diabetic Retinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eye Clinic Medic Zuljan Jukic (Other)
Collaborators: Clinical Hospital Center, Split (Other); University of Zagreb (Other)
Responsible Party: Principal Investigator, Ljubo Znaor, Ophthalmologist, Clinical Hospital Center, Split
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MZJ-2106
Record Dates: First submitted 2012-09-23; First posted 2012-09-27 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Macular Edema; Cataract; Diabetic Retinopathy
Keywords: Macular edema; Cataract; Diabetic retinopathy; Anti-inflammatory agents,Non-steroidal
MeSH Terms: conditions — Macular Edema; Cataract; Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diclofenac (Experimental): Patients with diabetic retinopathy having preoperative treatment with diclofenac
  Interventions: Drug: Perioperative Diclofenac eye-drops administration
- Placebo (Placebo Comparator): Control group having placebo treatment
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Perioperative Diclofenac eye-drops administration
  Arms: Diclofenac
Drug: placebo
  Arms: Placebo

SUMMARY:
Diabetes has many negative effects on patients' general health. Among many other consequences it speeds up the cataract formation and that is why diabetic patients need cataract surgery very often. The known side effect of cataract surgery even in otherwise healthy patients is postoperative edema of the back of the eye (what causes decrease of vision), which has greater incidence especially in patients who have diabetic eye problems. The cause of that might be the intraocular inflammation which was previously demonstrated to be significantly more prominent in patients with untreated diabetic eye problems. Therefore we will examine if the 7 day use of anti-inflammatory eye drops prior to the cataract surgery prevent the formation of the edema of the back of the eye.

ELIGIBILITY:
Inclusion Criteria:

* presence of nonproliferative diabetic retinopathy
* presence of the cataract (LOCS 2-3)

Exclusion Criteria:

* other chronic or acute eye diseases
* hypersensitivity to any component of the diclofenac eye-drops patients on oral anticoagulant therapy
* allergy to salycilates

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-10; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change of Central Macular Thickness | -7, 0, 1, 7, 30, 90 days after the cataract surger
  The central macular thickness will be measured with OCT machine.

SECONDARY OUTCOMES:
progression of diabetic retinopathy | -7 and 90 days after cataract surgery
  The grade of diabetic retinopathy will be assessed on fundus photographies according to ETDRS criteria
IL-12 concentration | immediately before cataract surgery
  The IL-12 concentration will be measured in the sample of humour aqueous taken at the beginning of cataract surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ljubo Znaor, MD PhD, Principal Investigator — Clinical Hospital Center, Split
Locations (1):
- Poliklinika Medic Zuljan Jukić, Split, Croatia